CLINICAL TRIAL: NCT05371197
Title: Envafolimab as Neoadjuvant Immuntherapy in Resectable Local Advanced dMMR/MSI-H Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Vice-president of Third Affiliated Hospital, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENCC
Record Dates: First submitted 2021-11-29; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Mismatch Repair-deficient (dMMR); Microsatellite Instability-high (MSI-H); Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — Neoadjuvant Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 inhibitor (Experimental): Neoadjuvant therapy with PD-L1 inhibitor (Envafolimab)
  Interventions: Drug: Neoadjuvant therapy with PD-L1 inhibitor

INTERVENTIONS:
Drug: Neoadjuvant therapy with PD-L1 inhibitor — Neoadjuvant therapy with PD-L1 inhibitor (Envafolimab), 300mg, Q3W for 4 cycles

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignant tumours of human beings. Mismatch Repair-deficient (dMMR)/ Microsatellite Instability-high (MSI-H) CRC is a specific subtype of CRC, which accounts for approximately 15% of all CRC patients, and can not benefit from 5-fluorouracil (5-FU) adjuvant chemotherapy. Once patients have distant metastases, they are not sensitive to traditional palliative chemotherapy, and thus lead to much worse prognosis than that of mismatch repair-proficient (pMMR)/ microsatellite stability (MSS). A phase II clinical study of anti-PD-1 immunotherapy based on mismatch repair (MMR) status published in "N Engl J Med" showed that the objective response rate (ORR) of advanced colorectal cancer patients with dMMR received anti-PD-1 is 40%, and a longer response time can be obtained compared to conventional chemotherapy. Another study (ClinicalTrials.gov, NCT03926338) which investigating the effect of neoadjuvant PD-1 blockade with toripalimab, with or without celecoxib, on mismatch repair-deficient or microsatellite instability-high, locally advanced, colorectal cancer. The result revealed that all 34 patients had an R0 resection. 15 of 17 patients (88%) in the toripalimab plus celecoxib group and 11 of 17 patients (65%) in the toripalimab monotherapy group had a pathological complete response.

In theory, anti-PD-L1 drugs should have fewer immune side-effects than anti-PD-1 drugs. However, there are no reports of anti-PD-L1 neoadjuvant therapy for the dMMR/MSI-H colorectal cancer. Therefore, the aim of this study was to investigate the efficacy and safety of anti-PD-L1 monoclonal antibody (Envafolimab) as neoadjuvant immuntherapy for resectable local advanced colorectal cancer patient with the dMMR/MSI-H.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum.
3. Tumor tissues were identified as mismatch repair-deficient (dMMR) by immunohistochemistry (IHC) method or microsatellite instability-high (MSI-H) by polymerase chain reaction (PCR).
4. Male or female subjects > 18 years < 70 of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Determined CT or MRI scans (done within 14 days of registration) of the chest, abdomen and pelvis: locally advanced (cT3-4 or cN1-2 [with the definition of a clinically positive lymph node being any node ≥ 1.0 cm]).
7. Non complicated primary tumor (obstruction, perforation, bleeding).
8. No previous any systemic anticancer therapy for colorectal cancer disease or radiologic evaluation of tumor regression < 20% or unacceptable toxic effects during neoadjuvant chemotherapy.
9. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment.

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.
2. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
3. Heart failure grade III/IV (NYHA-classification).
4. Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
5. Subjects with known allergy to the study drugs or to any of its excipients.
6. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
7. Breast- feeding or pregnant women
8. Lack of effective contraception.
9. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.
10. With any distant metastasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates | 1 year
  Proportion of patients experiencing a pCR to perioperative PD-L1 antibody

SECONDARY OUTCOMES:
Major pathological response rates | 1 year
  The proportion of patients experiencing a major pathological response to perioperative PD-L1 antibody
R0 resection rates | 1 year
  The proportion of patients experiencing a R0 resection after perioperative treatment with PD-L1 antibody
Disease-free survival (DFS) | 3 years
  Defined as the time from randomization to relapse, metastasis or death from any cause
Overall survival (OS) | 5 years
  Defined as the time from randomization to death from any cause
Drug Safety | 1 year
  Assessed by evaluation of treatment-related adverse events
Drug feasibility | 1 year
  Any treatment-related delays in the planned surgery of no more than 28 days after the last preoperative toripalimab dose

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided